CLINICAL TRIAL: NCT04396210
Title: Patients Perspectives on Discontinuation of Their Fertility Treatment Due to the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000247
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus; COVID; ART; Fertility Issues
MeSH Terms: conditions — Coronavirus Infections; Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Eligible patients will be selected electronically from our database and digital agenda. After selection, patients will be contacted via email to participate. Two reminders will be send in case the questionnaire is not filled out: a first reminder after one week, a second reminder after two weeks.

SUMMARY:
The COVID-19 pandemic brought new challenges to our nationwide healthcare system, with rapid escalation of the number of affected individuals over a handful of weeks. From March 13, a first set of measures was taken to minimise the spread of the virus, which largely impacted societal and economical daily life. A view days later, on March 17, the country was put in "lockdown" and all non-urgent medical treatments were cancelled or postponed. As recommended by the major scientific fertility societies, all non-ivf fertility treatments were discontinued abruptly, whereas started ivf stimulations were continued until oocyte aspiration, where after a freeze-all strategy was applied.

There is little information available for women aiming for pregnancy or embarking on assisted conception. Given the modelling of the pandemic, including the time to peak and subsequent tail, considerable delays in conception to substantially attenuate risk may be required, which will inevitably impact patients wellbeing and overall success rates.

A questionnaire was developed to explore patients perspectives on different aspects of their fertility treatment during the COVID-19 pandemic.

The questionnaire contains the following sections:

* demographic variables;
* questions regarding the fertility history of the respondent;
* questions regarding the impact of fertility treatment cancellation / postponing fertility treatment during COVID-19 on their life, psychological wellbeing and relationship;
* questions regarding continuing medical treatment on their own, or seeking treatment elsewhere;
* questions regarding the satisfaction of measures taken by their fertility center regarding the COVID-19 pandemic;
* questions regarding expectations of further treatments, with focus on safety issues related to the COVID-19 pandemic.

Eligible patients will be selected electronically from our database and digital agenda. After selection, patients will be contacted via email to participate. Two reminders will be send in case the questionnaire is not filled out: a first reminder after one week, a second reminder after two weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients that did not start a fertility treatment yet ("intake group") OR;
* patients for which a treatment plan was made, but treatment was postponed ("before treatment") OR;
* patients who were undergoing a non-inf treatment cycle (ovulation-induction (OI), intra-uterine insemination (IUI)) and whose cycle was cancelled after starting the treatment cycle ("non-ivf treatment group") OR;
* patients who were undergoing a cryo cycle and whose cycle was cancelled after starting the treatment cycle ("cryo treatment group") OR;
* patients who were undergoing an IVF treatment cycle and for whom fresh embryo transfer was cancelled (freeze-all group).

Exclusion Criteria:

* Language other than Dutch

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients whose fertility treatment was discontinued abruptly due to the COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Patients perspectives on the abruptly discontinuation of their fertility treatment by using a questionnaire | During the COVID-19 pandemic, from March 2020 till June 2020
Patients reproductive behaviour by using a questionnaire | During the COVID-19 pandemic, from March 2020 till June 2020
Patients views on resuming fertility treatment by using a questionnaire | During the COVID-19 pandemic, from March 2020 till June 2020

CONTACTS AND LOCATIONS:
Overall Officials: Frauke Vanden Meerschaut, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No